CLINICAL TRIAL: NCT01635010
Title: Obstructive Sleep Apnea in the Absence of Metabolic Syndrome: Pulse Wave Velocity, Inflammatory and Oxidative Stress Markers
Brief Title: Obstructive Sleep Apnea in the Absence of Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Associação Fundo de Incentivo à Pesquisa (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Daniela Kuguimoto Andaku Olenscki, Doctoral researcher, Associação Fundo de Incentivo à Pesquisa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASSIMVOP012
Record Dates: First submitted 2012-06-29; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; inflammation; oxidative stress; arterial stiffness
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Obstructive sleep apnea (Experimental)
  Interventions: Procedure: continuous positive airway pressure (CPAP)

INTERVENTIONS:
Procedure: continuous positive airway pressure (CPAP) — CPAP pressure is individually prescript according to polysomnography for CPAP titration
  Arms: Obstructive sleep apnea

SUMMARY:
Obstructive Sleep Apnea (OSA) is commonly associated with factors that increase cardiovascular risk, including Metabolic Syndrome (MS). There is a lack of well-controlled clinical studies investigating the independent effects of OSA in the development of cardiovascular disease, especially evaluating jointly mechanisms involved in these disorders such as inflammatory response, oxidative stress and vascular changes. The investigators hypothesized that in the absence of MetS, the mechanisms involved on cardiovascular consequences in OSA patients would be less important.

The purpose of this study is to analyze the effects of OSA in the absence of MS, on inflammatory, oxidative stress and vascular markers; to verify the influence of excessive daytime sleepiness (EDS) on the same parameters; and additionally verify the effects of nasal continuous positive airway pressure (nCPAP)in theses parameters.

ELIGIBILITY:
Inclusion Criteria:

* male subjects
* apnea-hypopnea index > 15/h (OSA group)
* apnea-hypopnea index < 5/h (control group)

Exclusion Criteria:

* body mass index (BMI) > 30 kg/m2
* age > 60 years
* chronic obstructive pulmonary disease
* cardiac diseases
* diabetes mellitus
* metabolic syndrome according to modified National Cholesterol Education Program Adult Treatment Panel III criteria
* previous OSA treatment

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Inflammatory marker (high sensitive C-reactive protein) | 3 months
Oxidative stress marker (homocysteine, cysteine and paraoxonase-1 activity) | 3 months
Arterial stiffness (pulse wave velocity) | 3 months
Angiotensin converting enzyme activity | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniela K. Andaku, MSc, Principal Investigator — Associação Fundo de Incentivo à Pesquisa; Sônia M. Togeiro, PhD, Study Chair — Associação Fundo de Incentivo à Pesquisa; Vânia D'Almeida, PhD, Study Chair — Associação Fundo de Incentivo à Pesquisa
Locations (1):
- Associação Fundo de Incentivo à Pesquisa, São Paulo, São Paulo, Brazil